CLINICAL TRIAL: NCT05393739
Title: Effect of Transcranial Magnetic Stimulation on Visual Functions of Adult Amblyopia: a Preliminary Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202106139DINC
Record Dates: First submitted 2022-05-02; First posted 2022-05-26 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Amblyopia
Keywords: Transcranial magnetic stimulation; Amblyopia; Neuroplasticity
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intermittent theta burst (Experimental): The total TBS time is about 1 to 3 minutes and the subjects have to look at at a visual stimulus on a computer monitor while receiving TBS and continue the visual training until 20 minutes after the treatment. In iTBS group, the subjects look at the visual stimulus with amblyopic eye while in cTBS group, subjects look at visual stimulus with non-amblyopic eye. The subjects will receive three times of stimulations in one week. The visual function evaluation includes BCVA, contrast sensitivity and stereoacuity. Visual functions will be evaluated right after TBS session (t1). Participant will receive same type of treatment for another 2 times within one week followed by visual function tests (t2). To evaluate the long-term effect, participants will be followed for another visual function tests (t3) after 2 weeks.
  Interventions: Device: Theta burst transcranial magnetic stimulation (TBS) procedure
- Continuous theta burst (Experimental): The total TBS time is about 1 to 3 minutes and the subjects have to look at at a visual stimulus on a computer monitor while receiving TBS and continue the visual training until 20 minutes after the treatment. In iTBS group, the subjects look at the visual stimulus with amblyopic eye while in cTBS group, subjects look at visual stimulus with non-amblyopic eye. The subjects will receive three times of stimulations in one week. The visual function evaluation includes BCVA, contrast sensitivity and stereoacuity. Visual functions will be evaluated right after TBS session (t1). Participant will receive same type of treatment for another 2 times within one week followed by visual function tests (t2). To evaluate the long-term effect, participants will be followed for another visual function tests (t3) after 2 weeks.
  Interventions: Device: Theta burst transcranial magnetic stimulation (TBS) procedure
- Sham theta burst (Sham Comparator): The stimulus intensity in sham group is about half of that in iTBS/cTBS groups, and the subjects receive a placebo stimulation with the coil orientation tilted to 90°. The visual function evaluation includes BCVA, contrast sensitivity and stereoacuity. Visual functions will be evaluated right after TBS session (t1). Participant will receive same type of treatment for another 2 times within one week followed by visual function tests (t2). To evaluate the long-term effect, participants will be followed for another visual function tests (t3) after 2 weeks.
  Interventions: Device: Theta burst transcranial magnetic stimulation (TBS) procedure

INTERVENTIONS:
Device: Theta burst transcranial magnetic stimulation (TBS) procedure — The procedure includes determining the specific occipital point at which place the stimulation coil; this corresponds to the area where magnetic stimulation is most capable of inducing phosphenes or transient visual phenomena. The phosphenes are directly induced by stimulation of the visual cortex and their presence indicates that the magnetic stimulation is in the correct location. The subjects would wear a personalized swimming cap with the determined area for stimulation marked on it. The major differences between iTBS and cTBS are the frequency and interval of stimulus.

SUMMARY:
Amblyopia, with a prevalence rates of 3% in adult population, is a common cause of vision impairment. It is characterized by impaired vision in one or both eyes because of disruption of normal visual stimuli and underdevelopment of the visual cortex, leads to lifelong visual deficits affecting both monocular and binocular visual function. Common causes of amblyopia include refraction error, anisometropia, strabismus and visual deprivation arising from ptosis or congenital cataract. Our previous studies had shed light on the relationship between abnormal early visual experience, and development of later amblyopia and possible neural developmental disorders. Functional recovery is difficult when neuroplasticity slows down at the end of the critical period. To date, there is no established effective treatment for adult amblyopia.

Repetitive transcranial magnetic stimulation (rTMS) is one of the non-invasive stimulations had been used widely as a research tool to understand the brain functions and an established treatment modality in neuropsychiatric diseases. Theta burst stimulation (TBS) is a newer form of rTMS protocol which have a major advantage over traditional rTMS in their reduced administration duration and allowing stimulation at significantly lower intensities to attain comparable effects. TBS had been demonstrated to able to improve functions in participants with visual disorders. However, studies of its use on adult amblyopia are scarce. Due to lack of efficient treatment at present, it is of scientific significance to conduct placebo-controlled experiments on this topic. Investigators will evaluate the effect of three regimens of TBS (intermittent, continuous and sham), after one session and accumulative sessions, on visual functions of amblyopia adults shortly after treatment and 2 weeks later (lasting effect), in order to evaluate its potential role in amblyopia and find out the best paradigm for amblyopia treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult amblyopia participants, aged 20-50 years old.
2. Based on inclusion criteria, there was a minimum of 2 lines difference in BCVA between the 2 eyes.
3. An amblyogenic factor and history of amblyopia treatment was recorded

Exclusion Criteria:

1. Unstable vital sign
2. History of brain injury and/or head trauma
3. Neurological and psychiatric disease
4. Seizures or family history of seizure
5. Pregnancy
6. Uncontrolled migraine or the presence of metallic implants or shunt in the head or torso
7. Wide region of ischemic cicatrix, multiple sclerosis, taking tricycle antidepressants,
8. Analgesics or any drugs may decrease the threshold for inducing seizure
9. Experienced sleep disorders during the rTMS treatment
10. Severe alcoholism or taking seizure drugs
11. Severe heart diseases or uncontrollable migraine caused by high intracranial pressure

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective | 1 month for each participant
  Change from baseline best corrected visual acuity: distance visual acuity measured for each eye at a distance of 6 m. Visual acuity scored letter-by-letter instead and lonarithm of the minimum angle of resolution (logMAR) scores were recored.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Hsun Tsai, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei County, Taiwan